CLINICAL TRIAL: NCT06099431
Title: Reliability of a 2.3mm Mandibular Reconstruction Bone Plate in Mandibular Bone Preservation
Brief Title: Mandibular Reconstruction Bone Plate
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed Kamal Eid Allam, Associate professor, Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A23030123
Record Dates: First submitted 2023-10-09; First posted 2023-10-25 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-02

CONDITIONS: Mandible Tumor
Keywords: Reconstruction; bone plate; Mandible
MeSH Terms: conditions — Mandibular Neoplasms | interventions — Plastic Surgery Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Surgery/Device (Other): Mandibular marginal resection and reconstruction using a mandibular osteosynthesis a 2.3mm reconstruction bone plate
  Interventions: Procedure: Mandibular marginal resection and reconstruction; Device: mandibular osteosynthesis a 2.3mm reconstruction bone plate

INTERVENTIONS:
Procedure: Mandibular marginal resection and reconstruction — Intraoral buccal and lingual incisions 2-3 mm away from the free gingival margins were carried out around the teeth to be included in the resection. The osteotomy lines were marked using a long shank surgical tapered fissure bur. The osteotomies completed and the resected segment was removed.
Device: mandibular osteosynthesis a 2.3mm reconstruction bone plate — a 2.3 mm reconstruction bone plate was then fit in place and fixed to both the proximal and distal segments

SUMMARY:
The purpose of this study is to evaluate the reliability of using mandibular osteosynthesis a 2.3mm reconstruction bone plate in the maintenance of the space, contour, and mandibular bone preservation during marginal mandibular resection.

DETAILED DESCRIPTION:
This prospective study included 16 patients (n=16) suffering from presence of mandibular central benign lesions indicated for marginal mandibular resection.

Patient history included personal data (name, age, sex, and occupation), date of lesion discovery, mode of growth (rapid or slow), and symptoms (e.g. pain and/or ipsilateral paresthesia of the lower lip).

Clinical examination included the site and extent of mandibular bony expansion and covering soft tissues (normal, ulcerated from indentation of opposing teeth, or scarred due to previous incisional biopsy).

Radiographical examination involved orthopantomography (OPG) and axial and coronal computed tomography (CT) scans to assess the lesion extensions.

All patients are operated under general anesthesia which was induced by intravenous access. Intubation is routinely performed in nasoendotracheal fashion.

Intraoral buccal and lingual incisions 2-3 mm away from the free gingival margins are carried out around the teeth to be included in the resection.

The plastic template is adapted to the buccal cortex of the mandible to aid in the final adaptation of a 2.3 mm reconstruction bone plate (Antonhib, Germany). The osteotomy lines are marked using a long shank surgical tapered fissure bur. a 2.3 mm reconstruction bone plate is then fit in place and fixed to both the proximal and distal segments then removed. The osteotomies completed and the resected segment is removed, and the reconstruction plate is then replaced by the aid of screw holes in both the proximal and distal segments. The intraoral wound is carefully closed in double layers using a combination of interrupted and horizontal mattress resorbable 3/0 sutures.

post operative follow up clinically regarding soft tissue healing, pain, infection, and plate exposure or plate fracture. Radiographically, Panoramic radiographs are taken immediately and axial and coronal computed tomography at six months post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from presence of mandibular central benign lesions indicated for marginal mandibular resection

Exclusion Criteria:

* systemic disease affect primary wound healing malignancy

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 16 (Estimated)
Dates: Start 2022-12-22 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Degree of pain | 1 month
  The degree of pain is determined during the follow up periods according the scale of Kerkmanov and Nordenram , Mild: require one tablet of analgesics three times/ day, Moderate: require two tablets of analgesics three times/ day, Severe: require injective analgesics.
Rate of inflammation | 1 month
  The wounds were inspected accurately post-operatively for detecting the proper healing using inflammation score scale, 0 no inflammation,1-3 mild inflammation, 4-7,moderate inflammation, 8-10 sever inflammation
Rate of Infection | 6 months
  using Infection score scale , mild infection which responds to antibiotics, only without the need for incision and drainage, moderate infection which needs for incision and drainage and severe infection which needs for incision and drainage in addition to hardware removal.

SECONDARY OUTCOMES:
Axial and coronal computed tomography | 6 month
  Degree of bone plate stability

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed K Allam, Ass prof, Principal Investigator — Tanta University
Locations (1):
- Tanta University, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No